CLINICAL TRIAL: NCT02553239
Title: CoolLoop Paroxysmal Atrial Fibrillation
Acronym: CoolLoop PAF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient patient recruitment
Sponsor: afreeze GmbH (Other)
Collaborators: Accovion GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CoolLoop PAF
Record Dates: First submitted 2015-09-14; First posted 2015-09-17 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation (Paroxysmal); Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Diseases; Pathologic Processes
Keywords: Atrial Fibrillation; Paroxysmal; Cryoablation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Diseases; Pathologic Processes | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryoablation (Experimental): Cryoablation with the CoolLoop® catheter
  Interventions: Device: CoolLoop®

INTERVENTIONS:
Device: CoolLoop® — Cryoablation of Atrial Fibrillation Using the CoolLoop Cryoablation System
  Other Names: Cryoablation; CoolLoop cryoablation system

SUMMARY:
This clinical investigation evaluates the safety of cryoablation (sclerotherapy of muscle tissue of the heart by freezing) in paroxysmal atrial fibrillation with the newly developed CoolLoop® cryoablation catheter.

A further aim of the investigation is the evaluation of the efficacy and average duration of the applied procedure.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 70 years
* symptomatic paroxysmal Atrial fibrillation (AF)
* a minimum of three episodes of paroxysmal AF
* at least one episode of paroxysmal AF within the last 6 months documented by ECG
* signed and dated informed consent documented by the patient
* female subjects of childbearing potential can be included, if they: agree to use, and be able to comply with, effective contraception without interruption, from study enrollment, throughout hospitalization and until 12 weeks after catheter ablation

Exclusion Criteria:

* left atrial diameter > 50 mm in the short axis as assessed by transthoracic echocardiography
* advanced structural heart disease including

  * moderate-to-severe valvular stenosis or regurgitation,
  * previous valve replacement or valve repair,
  * congenital heart disease,
  * left ventricular ejection fraction < 45% during sinus rhythm,
  * congestive heart failure New York Heart Association (NYHA) III or IV,
  * coronary artery bypass graft surgery within the last 3 months
* chronic obstructive pulmonary disease treated with beta-sympathomimetic drugs
* severe respiratory insufficiency
* known bleeding diathesis
* intolerance of Heparin and/or intolerance of oral anticoagulation
* previous AF ablation
* permanent pacemaker
* left atrial thrombus
* intramural or intracardiac thrombus or tumor, or other conditions that may result in difficulties advancing the CoolLoop® cryoablation catheter into the left atrium
* access to the vascular system via the right or left femoral vein is not possible
* transseptal puncture cannot be achieved due to a previous operation or intervention at the interatrial septum (e.g. closure of a patent foramen ovale or atrial septal defect)
* contraindication for transesophageal echocardiography or fluoroscopy
* impaired renal function (glomerular filtration rate <30 ml/min.)
* history or increased risk of intracranial hemorrhage
* history of cerebral ischemic stroke or transient ischemic cerebral attacks within the last 180 days prior to enrolment
* severe comorbidity
* hyperthyreosis
* any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he / she were to participate in the study or confound the ability to interpret data from the study
* any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the Informed Consent Form
* pregnant or lactating females
* other severe conditions, which makes the patient unsuitable to participate in the study, as judged by the Investigator
* live-expectancy < 1 year
* the patient is active in another clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Safety of catheter ablation using the CoolLoop® cryoablation catheter determined by the number of patients with device-, or procedure-related serious adverse events. | 12 months follow-up period

SECONDARY OUTCOMES:
Measurement of freedom from Atrial Fibrillation (AF) episodes following left atrial catheter ablation using the CoolLoop cryoablation catheter. | from 3 to 12 months after catheter ablation
  Number of patients without AF episodes, determined by continuous ECG recording for 7 days at 1 year after treatment.
Assessment of acute efficacy of catheter ablation defined by Pulmonary Vein (PV) Isolation. | from start to end of ablation procedure
  Acute efficacy is defined as the electrical isolation in ≥ 3 PVs at the end of the intervention. Estimated timeframe 360 minutes (average).
Assessment of the CoolLoop catheter procedure time | from start to end of ablation procedure
  Estimated timeframe 360 minutes (average).
Assessment of the CoolLoop fluoroscopy time | from start to end of ablation procedure
  Estimated timeframe 360 minutes (average).
Assessment of the CoolLoop cryoablation time | from start to end of ablation procedure
  Cryoablation time is specified as the cumulative "total freeze time" during treatment. Estimated timeframe 360 minutes (average).
Assessment of serious and non-serious Adverse Events (SAEs/AEs) | 12 months follow-up period
  Number of patients with SAEs and AEs

CONTACTS AND LOCATIONS:
Overall Officials: Karoline Etschmaier, PhD, Study Director — afreeze GmbH
Locations (4):
- Austria (2):
  - Medical University Innsbruck, Innsbruck, Tyrol
  - Allgemeines Krankenhaus der Stadt Linz, Linz, Upper Austria
- Klinik für Kardiologie, Bad Oeynhausen, North Rhine-Westphalia, Germany
- UniversitätsSpital Zuerich, Zurich, Switzerland